CLINICAL TRIAL: NCT01130610
Title: Pre-anesthetic Evaluation and Cost Reduction Perioperative
Brief Title: Pre-anesthetic Evaluation and Cost Reduction
Status: Completed | Type: Observational
Sponsor: Santa Casa de Misericórdia de Belo Horizonte (Other)
Responsible Party: Magda Lourenço Fernandes, Santa Casa de Misericórdia de Belo Horizonte
Other Study IDs: CEP 089/2009
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Surgical Procedures; Anesthesia
Keywords: preoperative period; preoperative care; anesthesia; program evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study conducted in large Brazilian hospital, with the main objective of evaluating the impact of pre-anesthetic in reducing costs related to the preoperative preparation of patients admitted to undergo surgery or diagnostic procedures under anesthesia.

DETAILED DESCRIPTION:
The pre-anesthetic evaluation is essential in the care of surgical patients. Among its benefits stands the reduction of costs related to preoperative preparation. However, most studies evaluating costs was performed in hospitals abroad, whose reality does not always apply to our environment. The aim of this study is to compare the costs of preoperative evaluation performed by the surgeon (conventional tillage), with the cost of preparation performed by the anesthesiologist (pre-anesthetic evaluation). Two hundred patients scheduled for surgical or diagnostic procedures under anesthesia form included in the study. After admission patients were assessed by physician anesthesiologists. In Form 1 (conventional tillage), it was noted tests or specialist consultations made in the preoperative period. In Form 2 (pre-anesthetic evaluation) was noted comorbidities, physical examination and complementary examinations given in accordance with the guidelines adopted by the Anesthesiology Department of the institution. Form data were compared with a data form 2. Besides the costs, we compared the number of tests considered unnecessary and disagreements in the classification of physical status according to the American Society Anesthesiology (ASA).

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of one year and admitted for surgery or diagnostic procedures under anesthesia
* patient did not undergo pre-anesthetic evaluation prior to admission to hospital

Exclusion Criteria:

* Emergency surgery
* Major surgery with hospitalization on a date prior to the operation

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to the institution to undergo elective surgery or diagnostic procedures with anesthesia.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa Márcia, graduate, Study Director — Santa Casa de Misericórdia de Belo Horizonte; Magda Fernandes, Master, Principal Investigator — Santa Casa de Misericórdia de Belo Horizonte
Locations (1):
- Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Power LM, Thackray NM. Reduction of preoperative investigations with the introduction of an anaesthetist-led preoperative assessment clinic. Anaesth Intensive Care. 1999 Oct;27(5):481-8. doi: 10.1177/0310057X9902700508. PMID 10520388
- [Result] Fischer SP. Development and effectiveness of an anesthesia preoperative evaluation clinic in a teaching hospital. Anesthesiology. 1996 Jul;85(1):196-206. doi: 10.1097/00000542-199607000-00025. No abstract available. PMID 8694365
- [Result] Pasternak LR. Preoperative laboratory testing: general issues and considerations. Anesthesiol Clin North Am. 2004 Mar;22(1):13-25. doi: 10.1016/S0889-8537(03)00115-9. PMID 15109688